CLINICAL TRIAL: NCT01306643
Title: Single-agent Idelalisib for Previously Treated Low-grade Lymphoma: A Phase 1/2 Study of Safety, Efficacy, and Flow-cytometric Assessment of Tumor-cell Signaling Events
Brief Title: Safety and Efficacy Study of Idelalisib (GS-1101, CAL-101) in Patients With Previously Treated Low-grade Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101-10
Record Dates: First submitted 2011-02-25; First posted 2011-03-02 (Estimated); Results first posted 2016-12-21 (Estimated); Last update posted 2018-11-19 (Actual); Status verified 2016-10

CONDITIONS: Indolent Non-Hodgkin's Lymphoma; Follicular Lymphoma; Small Lymphocytic Lymphoma; Marginal Zone Lymphoma
Keywords: Indolent Non-Hodgkin's Lymphoma; Non-Hodgkin Lymphoma; iNHL; NHL; CAL-101; PI3K; Phosphatidylinositol 3-kinase; Follicular Lymphoma (FL); Small Lymphocytic Lymphoma (SLL); Marginal Zone Lymphoma (MZL)
MeSH Terms: conditions — Lymphoma, Follicular; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Non-Hodgkin | interventions — idelalisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Idelalisib (Experimental)
  Interventions: Drug: Idelalisib

INTERVENTIONS:
Drug: Idelalisib — Tablet(s) administered orally twice daily
  Other Names: GS-1101; CAL-101; Zydelig®

SUMMARY:
The primary objectives of this study is to evaluate the safety and efficacy of idelalisib (GS-1101, CAL-101) in participants with previously treated indolent non-Hodgkin lymphoma (iNHL).

Eligible patients will initiate oral therapy with idelalisib at a starting dose of 150 mg twice per day. Treatment with idelalisib can continue in compliant participants for up to twelve 28-day cycles of idelalisib. Participants who appear to be benefiting from treatment at the completion of 12 cycles of treatment with idelalisib may be eligible for participation in a long-term safety extension study of idelalisib.

ELIGIBILITY:
Inclusion Criteria:

* Previously treated relapsed or refractory B-cell iNHL
* Provide written informed consent

Exclusion Criteria:

* Pregnant or nursing
* Active, serious infection requiring systemic therapy
* Positive test for HIV antibodies
* Active hepatitis B or C viral infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (2):
- United States (2):
  - Stanford Cancer Center, Palo Alto, California
  - Mount Sinai School of Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 2 study sites in the United States. The first participant was screened on 22 February 2011. The last study visit occurred on 24 August 2015.
Pre-assignment Details: 24 participants were screened.
Groups:
- Idelalisib: Idelalisib 150 mg tablet(s) administered orally twice daily for a maximum of twelve 28-day cycles
Period: Overall Study
Arm/Group | Idelalisib
Started | 18
Completed | 5 (Completed Study was defined as participants who completed through Cycle 12 (Week 48) per protocol.)
Not Completed | 13
Not completed — Adverse Event | 5
Not completed — Disease Progression | 7
Not completed — Other: Change in Eligibility Status | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) Analysis Set: all enrolled participants who received at least 1 dose of idelalisib.
Arm/Group | Idelalisib
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 10
Diagnosis [Number; unit: participants]
  Follicular lymphoma | 10
  Marginal zone lymphoma | 3
  Small lymphocytic lymphoma | 4
  Missing | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Safety of Idelalisib
Description: The overall safety of idelalisib was assessed as the percentage of participants experiencing treatment-emergent adverse events (AEs; Serious AEs, Grade ≥ 3 AEs, AEs related to idelalisib, and AEs leading to discontinuation of idelalisib).
Time Frame: 30 days post last study treatment (up to 12 months)
Population: Intent-to-treat (ITT) Analysis Set: all enrolled participants who received at least 1 dose of idelalisib.
Measure: Number; unit: percentage of participants
Arm/Group | Idelalisib
Number analyzed (Participants) | 18
percentage of participants
  Any AE | 88.9
  Serious AE | 27.8
  Grade ≥ 3 AE | 55.6
  AE related to idelalisib | 83.3
  AE leading to permanent drug discontinuation | 27.8

2. Primary Outcome: Clinical Response: Overall Response Rate
Description: Participants were assessed for clinical response by appropriate imaging at the end of cycles 3, 6, 9, and 12.
  Overall response rate (ORR) was assessed based on standardized criteria (Cheson 2007), and was defined as the percentage of participants who achieved a complete response (CR) or partial response (PR) based on investigator assessment after the start of idelalisib treatment until progression or the end of study drug treatment.
  * CR was defined as the disappearance of all evidence of disease.
  * PR was defined the regression of measurable disease and no new sites.
Time Frame: Up to twelve 28-day cycles (maximum of 12 months)
Population: ITT Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Idelalisib
Number analyzed (Participants) | 18
percentage of participants | 44.4 [21.5 to 69.2]

3. Secondary Outcome: Flow Cytometric Measurement of Constitutive or Inducible Phosphorylation of Akt (at S473) and S6 Within Tumor B Cells
Time Frame: Up to twelve 28-day cycles (maximum of 12 months)
Population: Data are not available because the samples and analysis results (performed at the sites) could not be retrieved by Gilead.
Arm/Group | Idelalisib
Number analyzed (Participants) | 0

4. Secondary Outcome: Flow Cytometric Measurement of Tumoral and Peripheral Blood T and NK Cells
Time Frame: Up to twelve 28-day cycles (maximum of 12 months)
Population: as for outcome 3
Arm/Group | Idelalisib
Number analyzed (Participants) | 0

5. Secondary Outcome: Changes in Concentration of Peripheral Blood Chemokines and Cytokines
Time Frame: Up to twelve 28-day cycles (maximum of 12 months)
Population: as for outcome 3
Arm/Group | Idelalisib
Number analyzed (Participants) | 0

6. Secondary Outcome: Changes in Liver Imaging as Assessed by Magnetic Resonance Imaging (MRI) and Gadoxetic Acid (GD-EOB-DTPA) Contrast
Time Frame: Up to twelve 28-day cycles (maximum of 12 months)
Population: as for outcome 3
Arm/Group | Idelalisib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 30 days post last study treatment (up to 12 months)
Description: ITT Analysis Set
Arm/Group | Idelalisib
Serious Adverse Events (participants affected / at risk) | 5/18
Other Adverse Events (participants affected / at risk) | 15/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Idelalisib (N=18)
Atrial fibrillation (Cardiac disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Cellulitis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Transaminases increased (Investigations) | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 2
Renal failure (Renal and urinary disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Idelalisib (N=18)
Neutropenia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Atrial fibrillation (Cardiac disorders) | 1
Atrial tachycardia (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 2
Blepharospasm (Eye disorders) | 1
Chalazion (Eye disorders) | 1
Conjunctival hyperaemia (Eye disorders) | 1
Keratitis (Eye disorders) | 1
Photopsia (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 8
Flatulence (Gastrointestinal disorders) | 3
Gastrointestinal pain (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Lip discolouration (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 7
Oral pain (Gastrointestinal disorders) | 1
Painful defaecation (Gastrointestinal disorders) | 1
Paraesthesia oral (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 5
Asthenia (General disorders) | 2
Chest pain (General disorders) | 1
Chills (General disorders) | 2
Fatigue (General disorders) | 8
Influenza like illness (General disorders) | 2
Malaise (General disorders) | 2
Pain (General disorders) | 2
Pyrexia (General disorders) | 5
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Atypical pneumonia (Infections and infestations) | 1
Candida infection (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Hordeolum (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 4
Contusion (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 8
Aspartate aminotransferase increased (Investigations) | 8
Blood bilirubin increased (Investigations) | 2
Blood creatinine increased (Investigations) | 1
Blood phosphorus increased (Investigations) | 1
Blood uric acid increased (Investigations) | 1
Glomerular filtration rate decreased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Transaminases increased (Investigations) | 4
Weight decreased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Dysgeusia (Nervous system disorders) | 3
Headache (Nervous system disorders) | 4
Hypersomnia (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 2
Mental impairment (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Sinus headache (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 2
Confusional state (Psychiatric disorders) | 1
Emotional disorder (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 5
Chromaturia (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Nocturia (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Hypopnoea (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Exfoliative rash (Skin and subcutaneous tissue disorders) | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 5
Skin fissures (Skin and subcutaneous tissue disorders) | 1
Hot flush (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years